CLINICAL TRIAL: NCT00968799
Title: Hyperthermic Intraoperative Intraperitoneal Chemotherapy of Recurrent Ovarian Cancer - A Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor patient accrual
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Sascha Müller, Oberarzt, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGOV01
Record Dates: First submitted 2008-02-12; First posted 2009-08-31 (Estimated); Results first posted 2013-05-10 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Carcinoma
Keywords: Ovarian Neoplasms; Recurrence; Hyperthermia, Induced; Peritoneal Neoplasms; recurrent epithelial ovarian cancer; recurrent fallopian tube carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Ovarian Neoplasms; Recurrence; Hyperthermia; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Cytoreduction Surgical Procedures; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPEC treatment (Experimental): Cytoreduction
  Hyperthermic intraoperative intraperitoneal chemotherapy (HIPEC) with cisplatin
  Perfusion of the peritoneum with 42°C warm 25 mg/l cisplatin solution. Perfusion volume depends on body size (3 - 6 l).
  If cisplatin amount exceeds the equivalent of 62.5 mg/m² body surface, cisplatin is dosed by body surface (62.5 mg/m²)(safety margin).
  Perfusion is performed with the open or Coliseum technique for 90 min.
  Interventions: Procedure: Hyperthermic intraoperative intraperitoneal chemotherapy; Procedure: Cytoreduction; Drug: Cisplatin

INTERVENTIONS:
Procedure: Hyperthermic intraoperative intraperitoneal chemotherapy — Perfusion of the peritoneum with 42°C warm 25 mg/l cisplatin solution.
  Other Names: HIPEC
Procedure: Cytoreduction — Surgical removal of tumor nodules
  including resection of organs infested with tumor
Drug: Cisplatin — Cisplatin is applied as chemotherapy during surgery
  Other Names: cis-diamminedichloroplatinum(II); cisplatinum; CDDP; Platinol

SUMMARY:
Most studies performing hyperthermic intraoperative intraperitoneal chemotherapy dose the cytotoxic drugs according to the body surface (like 50 mg/m² cisplatin) in analogy to systemic, intravenous chemotherapy (usually using the same dose). Although there seems to be a correlation between body surface and blood volume, the pharmacodynamics of drugs dosed by the body surface is still highly variable and thus dosing on the body surface is increasingly considered controversial for systemic administration.

For hyperthermic intraoperative intraperitoneal chemotherapy dosing by the body surface makes even less sense, since the aim is the highest possible drug concentration in the peritoneum without undue local and systemic toxicity. Furthermore, most studies using intraoperative chemotherapy vary the volume of the perfusate according to the size of the patient. Since the amount of cytotoxic drug is already fixed by the dosing on the body surface (amount [mg] = dose [mg/m²] x body surface [m²]) the effective concentration (mg/l) in the perfusate can vary considerably between patients. On the other hand pharmacokinetic analyses have shown that reducing the concentration of the cytotoxic drug in the perfusate reduces the efficacy even if the amount of the drug remains the same.

In this study the safety of a new dosing regime will be evaluated. The concentration of cisplatin in the perfusate will be held constant independent of body weight or size to achieve the highest effectiveness of the chemotherapy. The primary endpoint is the safety of the treatment. All patients should be able to receive full dose systemic carboplatin chemotherapy after completion the trial treatment.

DETAILED DESCRIPTION:
Disease Background:

Between 1997 and 2001 the incidence of ovarian cancer in Switzerland was 15.8 per 100'000 women and ranks fifth among the cancer incidence in women. Nearly half of the patients die of the disease leading to a mortality rate of 7.7 per 100'000. Together with pancreatic cancer, ovarian cancer ranks fifth among cancer related deaths in women. The most common form of ovarian cancer is the epithelial ovarian cancer with an incidence of 91.1%. Thus, in the following the term ovarian cancer will refer solely to malignant epithelial ovarian cancer (78.6% of all ovarian cancers) excluding borderline or low malignancy epithelial ovarian tumors (12.5%).

Early stages of the disease (FIGO I - IIA) show practically no symptoms, thus 80% of ovarian cancers are diagnosed at later stages (FIGO IIB - IV), a main reason for the high mortality. Treatment for all stages are surgical removal of visible and resectable tumor nodules, ovaries, uterus, omentum, pelvic and paraaortic lymph nodes, in advanced stages tumor infested organs or organ parts have to be removed (=cytoreduction or debulking). Survival time strongly depends on the completeness of the cytoreduction. Surgery is followed by a chemotherapy of carboplatin and paclitaxel or carboplatin alone (except for the low risk FIGO stage IA, G1).

Published survival rates after therapy vary considerably and are mainly dependent on the stage of the tumor and the remaining tumor size (some tumor masses cannot be resected due to the proximity to vital organs like major blood vessels).

_____Stage______survival after 5 years

* FIGO I........76% - 93%
* FIGO II.......60% - 74%
* FIGO III......23% - 41%
* FIGO IV..........11%

(from J. S. Berek & N. F. Hacker, Practical Gynecologic Oncology 3ed. Philadelphia: Lippincott Williams & Wilkins, 2000, 504.)

Even with optimal debulking and adjuvant chemotherapy about 55% of all patients suffer from recurrent ovarian cancer which is considered essentially an incurable disease, since the response rate of a secondary treatment is 30% and the median survival is about 60 weeks.

Therapy background:

Hyperthermic intraoperative intraperitoneal chemotherapy (HIPEC)

Unless the tumor has already metastasized (FIGO IV) ovarian cancer tumor nodules are restricted to the peritoneal cavity. Since standard chemotherapy is applied intravenously the cytotoxic drugs can reach the cancer cells only by diffusion into the peritoneum or via the blood stream by the sometimes poor vascularisation of the tumor nodules. To improve the exposure of the tumor to the cytotoxic drugs clinical trials were performed to deliver the chemotherapy directly into the peritoneum (intraperitoneal chemotherapy). While this type of therapy shows very promising results, it also has some serious drawbacks: permanent catheters have to be implanted, even distribution of the instillate is difficult and sometimes linked with considerable discomfort for the patient.

Alternatively the intraperitoneal chemotherapy can be applied directly after the cytoreductive surgery (intraoperative intraperitoneal chemotherapy). Since the peritoneum is completely opened, the perfusate can easily reach all surfaces and the surgeon can facilitate the distribution by gentle agitation with his hands. Since the whole procedure is performed during the surgery under full anesthesia the patient does not have to suffer additional discomfort. While intraperitoneal chemotherapy can be applied repeatedly like conventional chemotherapy, the intraoperative chemotherapy can only be performed once. Thus, the effectiveness of the treatment should be as high as possible. This can be achieved by using the highest possible drug concentration and by increasing the temperature of the perfusate to approximately 42°C (hyperthermic intraoperative intraperitoneal chemotherapy). The rational for the hyperthermic treatment is several fold. First, it has been shown that some tumors can be killed by elevated temperatures alone. Second, the elevated temperatures increase the diffusion rate of the drugs into the tumor and thus the drug can penetrate deeper into the tumor nodules. Furthermore, elevated temperatures increase the cell membrane permeability and thus the uptake of the cytotoxic drugs by the tumor cells. Finally, with some cytotoxic drugs, like cisplatin, the cytotoxicity can be increased about 50 fold by a temperature increase from 37°C to 42°C in tissue culture models.

Rationale for performing the trial:

Most studies performing hyperthermic intraoperative intraperitoneal chemotherapy dose the cytotoxic drugs according to the body surface (like 50 mg/m² cisplatin) in analogy to systemic, intravenous chemotherapy (usually using the same dose). Although there seems to be a correlation between body surface and blood volume, the pharmacodynamics of drugs dosed by the body surface is still highly variable and thus dosing on the body surface is increasingly considered controversial for systemic administration. However, only very few drugs are dosed differently, e.g. carboplatin.

For hyperthermic intraoperative intraperitoneal chemotherapy dosing by the body surface makes even less sense, since the aim is the highest possible drug concentration in the peritoneum without undue local and systemic toxicity. Furthermore, most studies using intraoperative chemotherapy vary the volume of the perfusate according to the size of the patient. Since the amount of cytotoxic drug is already fixed by the dosing on the body surface (amount [mg] = dose [mg/m²] x body surface [m²]) the effective concentration (mg/l) in the perfusate can vary considerably between patients. On the other hand pharmacokinetic analyses have shown that reducing the concentration of the cytotoxic drug in the perfusate reduces the efficacy even if the amount of the drug remains the same.

In this study the safety of a new dosing regime will be evaluated. The concentration of cisplatin in the perfusate will be held constant independent of body weight or size to achieve the highest effectiveness of the chemotherapy. However, if the amount of cisplatin would exceed the equivalent of 62.5 mg/m² body surface, dosing would be again based on the body surface (62.5 mg/m²) for safety reasons.

The primary endpoint is the safety of the treatment. All patients should be able to receive full dose systemic carboplatin chemotherapy after completion the trial treatment.

Treatment plan:

Patients undergo cytoreductive surgery to remove all visible tumor nodules.

After the cytoreduction the hyperthermic intraoperative intraperitoneal chemotherapy is performed. For 90 min 42°C warm cisplatin solution (25 mg/l) is perfused through the peritoneum. Afterwards cisplatin will be removed by repeatedly rinsing the peritoneum with Ringer lactate solution. During the whole procedure the patient will receive a strong hydration according to a predefined protocol.

Cisplatin pharmacokinetics:

The concentration of platinum will be determined in perfusate, plasma and urine at various time points.

Various published pharmacokinetic models of cisplatin clearance will be tested with the data obtained. Furthermore, we want to test whether pharmacokinetic parameters might correlate with nephrotoxicity to allow a prediction of nephrotoxic events.

Translational research:

Tumor tissue removed during the cytoreduction will be used for various in vitro experiments:

* Histological examination for infiltrating lymphocytes and determination of the lymphocytes
* Determine the depth of platinum infiltration after treatment of the tumor nodules under various conditions with cisplatin (in vitro)
* Analysis of tumor cell biology after chemotherapy and heat treatment in vitro (protein phosphorylation, release of second messengers)

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed and recurrent epithelial ovarian carcinoma, fallopian tube carcinoma or primary peritoneal carcinoma requiring secondary debulking. Last chemotherapy of primary treatment was finished at least 6 months before.
* Patient must give written informed consent before registration
* WHO/ECOG performance status 0 - 1
* Age ≥18 years, ≤70 years
* Adequate hematological values: leukocytes ≥3x10^9/l, thrombocytes ≥100x10^9/l
* Adequate renal function. Obstructive hydronephrosis as a cause of "borderline" (30 - 45 ml/min) renal function should be investigated and treated prior to study entry.
* Patient compliance and geographic proximity allow proper staging and follow-up.
* FIGO III and IV

Exclusion Criteria:

* Primary diagnosis of epithelial ovarian cancer, or primary treatment completed less than 6 months ago.
* FIGO stage I + II
* Distant and current metastases
* WHO/ECOG performance status ≥2
* Inadequate hepatic function: bilirubin >1.5x ULN (upper limit normal range) or ASAT/ALAT >2.5x ULN or AP >5x ULN
* Psychiatric disorder precluding understanding of information of trial related topics or giving informed consent
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to trial entry
* Any serious underlying medical condition (at the judgment of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes)
* Known hypersensitivity to cisplatin
* Any concomitant drugs contraindicated for use with the trial drugs according to the Swissmedic-approved product information
* Dehydration
* Impaired hearing or symptomatic peripheral neuropathy: ≥grade II NCI-CTCAEv3
* Regular use of anti-epileptics

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Lüdin, MD, Principal Investigator — Cantonal Hospital St. Gallen, Department of Surgery
Locations (1):
- Department of Surgery, Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: overall recruitment was poor. study was terminated after 6 patients (of 27 scheduled)
Groups:
- HIPEC: Hyperthermic intraoperative intraperitoneal chemotherapy (HIPEC)
  Tumor nodules are removed surgically. If necessary infested organs like colon are resected (=cytoreduction).
  To destroy remaining tumor cells or invisible nodules the peritoneum is prefused with 42°C warm 25 mg/l cisplatin solution. Perfusion volume depends on body size (3 - 6 l).
  If cisplatin amount exceeds the equivalent of 62.5 mg/m² body surface, cisplatin is dosed by body surface (62.5 mg/m²)(safety margin).
  Perfusion is performed with the open or Coliseum technique for 90 min.
Period: Overall Study
Arm/Group | HIPEC
Started | 6
Completed | 4
Not Completed | 2
Not completed — Advanced disease, HIPEC not applicable | 2

BASELINE CHARACTERISTICS:
Groups:
- HIPEC: Hyperthermic intraoperative intraperitoneal chemotherapy (HIPEC)
Arm/Group | HIPEC
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 6

OUTCOME MEASURES:

1. Primary Outcome: Fitness for Systemic Chemotherapy
Description: Are patients fit to receive six courses of systemic carboplatin chemotherapy after completion of trial.
  If chemotherapy starts within 3 months after surgery and at least 4 courses could be administered, patient is considered fit.
  If chemotherapy is stopped early for reasons clearly unrelated to study treatment (e.g. platinum resistance), patient is also considered fit.
Time Frame: 3 months post operation
Measure: Number; unit: participants
Arm/Group | HIPEC
Number analyzed (Participants) | 4
participants | 4

2. Secondary Outcome: Nephrotoxicity
Description: glomerular filtration rate (GFR)
Time Frame: 6 weeks post operation
Measure: Number; unit: participants
Arm/Group | HIPEC
Number analyzed (Participants) | 4
participants
  no nephrotoxicity (normal GFR) | 2
  CTCAE grade 1 nephrotoxicity (by GFR) | 2

3. Secondary Outcome: Surgical Complications
Description: any serious surgical event (Dindo scale >= III (reoperation required) or CTCAE grade >=3)
Time Frame: 6 weeks post operation
Measure: Number; unit: participants
Arm/Group | HIPEC
Number analyzed (Participants) | 4
participants | 0

4. Secondary Outcome: Overall Survival
Time Frame: 5 years
Measure: Median (Full Range); unit: months
Arm/Group | HIPEC
Number analyzed (Participants) | 4
months | 26 [16 to 58]

5. Secondary Outcome: Pharmacokinetics
Description: data not analysed due to poor accrual
Time Frame: intraoperative and 1 week after surgery
Arm/Group | HIPEC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days post surgery
Arm/Group | HIPEC
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIPEC (N=4)
hypokalemia (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes